CLINICAL TRIAL: NCT03500133
Title: Non Randomized, Multicenter, Prospective Pediatric Hodgkin Lymphoma Treatment Trial Stratified According to Initial Risk Factors and Response to Chemotherapy, Reduced Cumulative Doses of Antineoplastic Agents and Radiotherapy.
Brief Title: Pediatric Hodgkin Lymphoma Treatment Trial With Low Cumulative Doses of Chemotherapy Agents and Reduced Radiation.
Acronym: LHGALOP2017
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital JP Garrahan (Other Government)
Responsible Party: Principal Investigator, Pedro Zubizarreta, MD, Hospital JP Garrahan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 991 Hodgkin Lymphoma GALOP2017
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Hodgkin's Disease
Keywords: Pediatric Hodgkin Lymphoma, therapy, reduced radiotherapy
MeSH Terms: interventions — ABVD protocol

STUDY DESIGN:
Intervention Model Description: Initial disease risk assignment defines three arms: low, intermediate and high risk. After early disease response assessment 7 Arms are defined, treated with more intense chemotherapy according to initial risk and therapy response. Finally radiotherapy is delivered only to patients who do not achieve complete remission after chemotherapy at late disease response assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group A (Experimental): Low risk with complete early response after two cycles of ABVD chemotherapy schedule. Only one more ABVD course is delivered.
  No radiotherapy if CR at the end of chemotherapy.
  Interventions: Radiation: No radiotherapy if CR at the end of chemotherapy.; Drug: Low risk with complete early response after two cycles of ABVD chemotherapy schedule. Only one more ABVD course is delivered.
- Group B (Experimental): Low risk with partial remission at early response assessment after two cycles of ABVD chemotherpay schedule. Two ABVD courses are delivered.
  No radiotherapy if CR at the end of chemotherapy
  Interventions: Radiation: No radiotherapy if CR at the end of chemotherapy.; Drug: Low risk with partial remission at early response assessment after two cycles of ABVD chemotherpay schedule. Two ABVD courses are delivered.
- Group B2 (Experimental): Low risk with partial remisssion after 4 cycles of ABVD chemotherapy schedule. Two ESHAP courses are delivered.
  No radiotherapy if CR at the end of chemotherapy. IN 30Gy RT in case of PR at the end of chemotherapy
  Interventions: Radiation: No radiotherapy if CR at the end of chemotherapy.; Drug: Low risk with partial remisssion after 4 cycles of ABVD chemotherapy schedule. Two ESHAP courses are delivered.; Radiation: IN 30Gy RT in case of PR at the end of chemotherapy
- Group C (Experimental): Intermediate risk with complete early response after two cycles of ABVD chemotherapy schedule. Three more ABVD courses are delivered.
  No radiotherapy if CR at the end of chemotherapy.
  Interventions: Radiation: No radiotherapy if CR at the end of chemotherapy.; Drug: Intermediate risk with complete early response after two cycles of ABVD chemotherapy schedule. Three more ABVD courses are delivered.
- Group D (Experimental): Intermediate risk with partial remission after two cycles of ABVD chemotherapy schedule. Four more chemotherapy courses are delivered alternating ESHAP and ABVD.
  No radiotherapy if CR at the end of chemotherapy. IN 30Gy RT in case of PR at the end of chemotherapy
  Interventions: Radiation: No radiotherapy if CR at the end of chemotherapy.; Radiation: IN 30Gy RT in case of PR at the end of chemotherapy; Drug: Intermediate risk with partial remission after two cycles of ABVD chemotherapy schedule. Four more chemotherapy courses are delivered alternating ESHAP and ABVD.
- Group E (Experimental): High risk with complete early response after 1 ABVD and 1 ESHAP courses. Four more chemotherapy courses are delivered alternating ESHAP and ABVD.
  No radiotherapy if CR at the end of chemotherapy
  Interventions: Radiation: No radiotherapy if CR at the end of chemotherapy.; Drug: High risk with complete early response after 1 ABVD and 1 ESHAP courses. Four more chemotherapy courses are delivered alternating ESHAP and ABVD.
- Group F (Experimental): High risk with partial remission after 1 ABVD and 1 ESHAP courses. Six more chemotherapy courses are delivered alternating ESHAP and ABVD.
  No radiotherapy if CR at the end of chemotherapy. IN 30Gy RT in case of PR at the end of chemotherapy
  Interventions: Radiation: No radiotherapy if CR at the end of chemotherapy.; Radiation: IN 30Gy RT in case of PR at the end of chemotherapy; Drug: High risk with partial remission after 1 ABVD and 1 ESHAP courses. Six more chemotherapy courses are delivered alternating ESHAP and ABVD.

INTERVENTIONS:
Radiation: No radiotherapy if CR at the end of chemotherapy. — Adapted chemotherapy without radiotherapy
Drug: Low risk with complete early response after two cycles of ABVD chemotherapy schedule. Only one more ABVD course is delivered. — Low risk with complete early response after two cycles of ABVD chemotherapy schedule. Only one more ABVD course is delivered.
  Arms: Group A
Drug: Low risk with partial remisssion after 4 cycles of ABVD chemotherapy schedule. Two ESHAP courses are delivered. — Low risk with partial remission at early response assessment after two cycles of ABVD chemotherpay schedule. Two ABVD courses are delivered.
  Arms: Group B2
Radiation: IN 30Gy RT in case of PR at the end of chemotherapy — Low risk with partial remisssion after 4 cycles of ABVD and 2 ESHAP courses: IN 30Gy RT
  Arms: Group B2; Group D; Group F
Drug: Intermediate risk with complete early response after two cycles of ABVD chemotherapy schedule. Three more ABVD courses are delivered. — Intermediate risk with complete early response after two cycles of ABVD chemotherapy schedule. Three more ABVD courses are delivered.
  Arms: Group C
Drug: Intermediate risk with partial remission after two cycles of ABVD chemotherapy schedule. Four more chemotherapy courses are delivered alternating ESHAP and ABVD. — Intermediate risk with partial remission after two cycles of ABVD chemotherapy schedule. Four more chemotherapy courses are delivered alternating ESHAP and ABVD.
  Arms: Group D
Drug: High risk with complete early response after 1 ABVD and 1 ESHAP courses. Four more chemotherapy courses are delivered alternating ESHAP and ABVD. — High risk with complete early response after 1 ABVD and 1 ESHAP courses. Four more chemotherapy courses are delivered alternating ESHAP and ABVD.
  Arms: Group E
Drug: High risk with partial remission after 1 ABVD and 1 ESHAP courses. Six more chemotherapy courses are delivered alternating ESHAP and ABVD. — High risk with partial remission after 1 ABVD and 1 ESHAP courses. Six more chemotherapy courses are delivered alternating ESHAP and ABVD.
  Arms: Group F
Drug: Low risk with partial remission at early response assessment after two cycles of ABVD chemotherpay schedule. Two ABVD courses are delivered. — Low risk with partial remission at early response assessment after two cycles of ABVD chemotherpay schedule. Two ABVD courses are delivered.
  Arms: Group B

SUMMARY:
This trial proposes a therapy for pediatric Hodgkin lymphoma with the objective of achieving high levels of long lasting complete remission with less risk of late effects.

Patients of both genders, between 2 and 18 years, with newly diagnosed classical Hodgkin lymphoma are admitted.

Initial staging provides stratification in three groups: low, intermediate and high risk. An initial set of two chemotherapy courses is administered to all cases after which a new disease assessment is performed. According to disease response a final therapy group is assigned. Rapid early responders benefit from less chemotherapy. At the end of chemotherapy, radiotherapy is delivered only to patients who do not achieve a complete response. Thus therapy is tailored to initial extension and disease responsiveness. Complete responders at the end of chemotherapy do not receive radiotherapy. Those who are in partial remission receive low dose (30Gy) involved node radiotherapy. Stable or progressive disease at any moment is assumed as a trial failure and new therapeutic strategies are offered to patients off protocol.

Chemotherapy is based upon regimes with well known effectiveness in Hodgkin lymphoma. (i.e. ABVD: doxorubicin, bleomycin, vinblastine and dacarbazine and ESHAP: Etoposide, methyl prednisolone, citarabine and cisplatin). The schedules are delivered with low cumulative drug doses and avoiding the use of toxic alkylating agents. Risks of secondary leukemia and infertility are thus minimized. Doxorubicin and bleomycin do not achieve cumulative doses that may expose to significant risk of heart or lung damage. Radiotherapy reduction avoids late radiation sequels.

This clinical study proposes a therapeutic approach based on chemotherapy that do not sum up high cumulative toxic doses. Therapy is tailored according to initial risk assessment and disease responsiveness. Those who achieve a complete response to chemotherapy do not receive additional radiotherapy, thus avoiding further late effects.

DETAILED DESCRIPTION:
This trial proposes a therapy for pediatric Hodgkin lymphoma with the objective of achieving high levels of long lasting complete remission with less risk of late effects.

Patients of both genders, between 2 and 18 years, with newly diagnosed classical Hodgkin lymphoma are admitted. An open surgical biopsy with histopatological diagnosis is preferred.

Initial staging provides stratification in three groups: low, intermediate and high risk. An initial set of two chemotherapy courses is administered to all cases after which an early disease response assessment is performed. According to disease response a final therapy group is assigned (7 arms).

Imaging with PET-CT and Deauville Score is preferred for initial and further disease assessment. Complete response is defined by volume reduction and metabolic remission. In case PET-CT is not available, CT and ultrasound with volume reduction standards to assess response may be used.

Rapid early responders who achieve complete remission (CR) benefit from less chemotherapy. Those who are in partial remission at the end of chemotherapy (late disease assessment) receive low dose (30Gy) involved node radiotherapy. At the end of chemotherapy, radiotherapy is delivered only to patients who do not achieve a CR. Thus, therapy is tailored according to initial extension and disease responsiveness. Complete responders at the end of chemotherapy do not receive radiotherapy. To avoid radiotherapy in the majority of cases constitutes a principal goal of this trial. Stable or progressive disease at any moment is assumed as a trial failure and new therapeutic strategies are offered to these patients off protocol.

Chemotherapy is based upon regimes with well known effectiveness in Hodgkin lymphoma. (i.e. ABVD: doxorubicin, bleomycin, vinblastine and dacarbazine and ESHAP: Etoposide, methyl prednisolone, citarabine and cisplatin).

Low risk arms (Arms A, B and B2) receive no more than 4 cycles of ABVD. Intermediate risk Arm C, 5 cycles of ABVD and Arm D 4 cycles of ABVD and 2 courses of ESHAP. High risk Arm E receives 3 cycles of ABVD and 3 Cycles of ESHAP, Arm F receives 4 courses of ABVD and 4 courses of ESHAP. The schedules are delivered projecting low cumulative drug doses and avoiding the use of toxic alkylating agents. Risks of secondary leukemia and infertility are thus minimized. Doxorubicin and bleomycin do not achieve cumulative doses that may expose to significant risk of heart or lung damage. Radiotherapy reduction avoids late radiation sequels.

Cardiac, lung , thyroid and any other toxic effects are prospectively assessed at onset and regularly during and after therapy.

The main event-free and overall survival proportions end points will be analyzed annually during the following 10 years after the last patient registration.

This clinical study proposes a therapeutic approach based on chemotherapy that do not sum up high cumulative toxic doses. Therapy is tailored according to initial risk assessment and disease responsiveness. Those who achieve a complete response after chemotherapy do not receive additional radiotherapy, thus avoiding further late effects.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of classical Hodgkin lymphoma.
* Normal renal, hepatic, pulmonary and metabolic function standards.
* Informed consent signed by patient and/or legal caretakers.

Exclusion Criteria:

* Lymphocyte predominant nodular Hodgkin lymphoma
* Any form of immunodeficiency before diagnosis. (primary immunodeficiencies, trasplant recipients or immunosuppressive therapies of any kind including corticoid therapies during 28 days before diagnosis).
* Pregnancy and breastfeeding period.
* Sexually active female patients who do not accept an effective contraceptive method during therapy.
* Positive HIV serology.
* Penfigus or hepatic ductopenia.
* Hodgkin lymphoma as a secondary malignant disease.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival | 3-10 years
  Event free survival probability (event= relapse or death)
Overall Survival | 3-10 years
  Overall survival probability (event= death)

SECONDARY OUTCOMES:
Acute, chronic or late toxic events | 0-10 years
  Number of patientsexperiencing treatment-related adverse effects and mortality according to CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital JP Garrahan, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Driscoll JJ, Rixe O. Overall survival: still the gold standard: why overall survival remains the definitive end point in cancer clinical trials. Cancer J. 2009 Sep-Oct;15(5):401-5. doi: 10.1097/PPO.0b013e3181bdc2e0. PMID 19826360
- [Background] Ellis LM, Bernstein DS, Voest EE, Berlin JD, Sargent D, Cortazar P, Garrett-Mayer E, Herbst RS, Lilenbaum RC, Sima C, Venook AP, Gonen M, Schilsky RL, Meropol NJ, Schnipper LE. American Society of Clinical Oncology perspective: Raising the bar for clinical trials by defining clinically meaningful outcomes. J Clin Oncol. 2014 Apr 20;32(12):1277-80. doi: 10.1200/JCO.2013.53.8009. Epub 2014 Mar 17. No abstract available. PMID 24638016
- [Background] Nachman JB, Sposto R, Herzog P, Gilchrist GS, Wolden SL, Thomson J, Kadin ME, Pattengale P, Davis PC, Hutchinson RJ, White K; Children's Cancer Group. Randomized comparison of low-dose involved-field radiotherapy and no radiotherapy for children with Hodgkin's disease who achieve a complete response to chemotherapy. J Clin Oncol. 2002 Sep 15;20(18):3765-71. doi: 10.1200/JCO.2002.12.007. PMID 12228196
- [Background] Wolden SL, Chen L, Kelly KM, Herzog P, Gilchrist GS, Thomson J, Sposto R, Kadin ME, Hutchinson RJ, Nachman J. Long-term results of CCG 5942: a randomized comparison of chemotherapy with and without radiotherapy for children with Hodgkin's lymphoma--a report from the Children's Oncology Group. J Clin Oncol. 2012 Sep 10;30(26):3174-80. doi: 10.1200/JCO.2011.41.1819. Epub 2012 May 29. PMID 22649136
- [Background] Dorffel W, Ruhl U, Luders H, Claviez A, Albrecht M, Bokkerink J, Holte H, Karlen J, Mann G, Marciniak H, Niggli F, Schmiegelow K, Schwarze EW, Potter R, Wickmann L, Schellong G. Treatment of children and adolescents with Hodgkin lymphoma without radiotherapy for patients in complete remission after chemotherapy: final results of the multinational trial GPOH-HD95. J Clin Oncol. 2013 Apr 20;31(12):1562-8. doi: 10.1200/JCO.2012.45.3266. Epub 2013 Mar 18. PMID 23509321
- [Background] Sackmann-Muriel F, Zubizarreta P, Gallo G, Scopinaro M, Alderete D, Alfaro E, Casak S, Chantada G, Felice MS, Quinteros R. Hodgkin disease in children: results of a prospective randomized trial in a single institution in Argentina. Med Pediatr Oncol. 1997 Dec;29(6):544-52. doi: 10.1002/(sici)1096-911x(199712)29:63.0.co;2-k. PMID 9324342
- [Background] Kelly KM, Sposto R, Hutchinson R, Massey V, McCarten K, Perkins S, Lones M, Villaluna D, Weiner M. BEACOPP chemotherapy is a highly effective regimen in children and adolescents with high-risk Hodgkin lymphoma: a report from the Children's Oncology Group. Blood. 2011 Mar 3;117(9):2596-603. doi: 10.1182/blood-2010-05-285379. Epub 2010 Nov 15. PMID 21079154
- [Background] Schwartz CL, Constine LS, Villaluna D, London WB, Hutchison RE, Sposto R, Lipshultz SE, Turner CS, deAlarcon PA, Chauvenet A. A risk-adapted, response-based approach using ABVE-PC for children and adolescents with intermediate- and high-risk Hodgkin lymphoma: the results of P9425. Blood. 2009 Sep 3;114(10):2051-9. doi: 10.1182/blood-2008-10-184143. Epub 2009 Jul 7. PMID 19584400
- [Background] Mauz-Korholz C, Hasenclever D, Dorffel W, Ruschke K, Pelz T, Voigt A, Stiefel M, Winkler M, Vilser C, Dieckmann K, Karlen J, Bergstrasser E, Fossa A, Mann G, Hummel M, Klapper W, Stein H, Vordermark D, Kluge R, Korholz D. Procarbazine-free OEPA-COPDAC chemotherapy in boys and standard OPPA-COPP in girls have comparable effectiveness in pediatric Hodgkin's lymphoma: the GPOH-HD-2002 study. J Clin Oncol. 2010 Aug 10;28(23):3680-6. doi: 10.1200/JCO.2009.26.9381. Epub 2010 Jul 12. PMID 20625128
- [Background] Zubizarreta PA, Alfaro E, Guitter M, Sanchez La Rosa C, Galluzzo ML, Millan N, Fiandrino F, Felice MS. Children and Adolescent Hodgkin Lymphoma in Argentina: Long-term Results After Combined ABVD and Restricted Radiotherapy. J Pediatr Hematol Oncol. 2017 Nov;39(8):602-608. doi: 10.1097/MPH.0000000000000943. PMID 28902084
- [Background] Mauz-Korholz C, Metzger ML, Kelly KM, Schwartz CL, Castellanos ME, Dieckmann K, Kluge R, Korholz D. Pediatric Hodgkin Lymphoma. J Clin Oncol. 2015 Sep 20;33(27):2975-85. doi: 10.1200/JCO.2014.59.4853. Epub 2015 Aug 24. PMID 26304892
- [Background] Johnson P, Federico M, Kirkwood A, Fossa A, Berkahn L, Carella A, d'Amore F, Enblad G, Franceschetto A, Fulham M, Luminari S, O'Doherty M, Patrick P, Roberts T, Sidra G, Stevens L, Smith P, Trotman J, Viney Z, Radford J, Barrington S. Adapted Treatment Guided by Interim PET-CT Scan in Advanced Hodgkin's Lymphoma. N Engl J Med. 2016 Jun 23;374(25):2419-29. doi: 10.1056/NEJMoa1510093. PMID 27332902
- [Background] Velasquez WS, McLaughlin P, Tucker S, Hagemeister FB, Swan F, Rodriguez MA, Romaguera J, Rubenstein E, Cabanillas F. ESHAP--an effective chemotherapy regimen in refractory and relapsing lymphoma: a 4-year follow-up study. J Clin Oncol. 1994 Jun;12(6):1169-76. doi: 10.1200/JCO.1994.12.6.1169. PMID 8201379
- [Background] Labrador J, Cabrero-Calvo M, Perez-Lopez E, Mateos MV, Vazquez L, Caballero MD, Garcia-Sanz R. ESHAP as salvage therapy for relapsed or refractory Hodgkin's lymphoma. Ann Hematol. 2014 Oct;93(10):1745-53. doi: 10.1007/s00277-014-2114-0. Epub 2014 May 27. PMID 24863692
- [Background] Furth C, Amthauer H, Hautzel H, Steffen IG, Ruf J, Schiefer J, Schonberger S, Henze G, Grandt R, Hundsdoerfer P, Dietlein M, Kobe C. Evaluation of interim PET response criteria in paediatric Hodgkin's lymphoma--results for dedicated assessment criteria in a blinded dual-centre read. Ann Oncol. 2011 May;22(5):1198-1203. doi: 10.1093/annonc/mdq557. Epub 2010 Oct 21. PMID 20966182
- [Background] Meignan M, Gallamini A, Itti E, Barrington S, Haioun C, Polliack A. Report on the Third International Workshop on Interim Positron Emission Tomography in Lymphoma held in Menton, France, 26-27 September 2011 and Menton 2011 consensus. Leuk Lymphoma. 2012 Oct;53(10):1876-81. doi: 10.3109/10428194.2012.677535. Epub 2012 Apr 23. PMID 22432519
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Engert A, Haverkamp H, Kobe C, Markova J, Renner C, Ho A, Zijlstra J, Kral Z, Fuchs M, Hallek M, Kanz L, Dohner H, Dorken B, Engel N, Topp M, Klutmann S, Amthauer H, Bockisch A, Kluge R, Kratochwil C, Schober O, Greil R, Andreesen R, Kneba M, Pfreundschuh M, Stein H, Eich HT, Muller RP, Dietlein M, Borchmann P, Diehl V; German Hodgkin Study Group; Swiss Group for Clinical Cancer Research; Arbeitsgemeinschaft Medikamentose Tumortherapie. Reduced-intensity chemotherapy and PET-guided radiotherapy in patients with advanced stage Hodgkin's lymphoma (HD15 trial): a randomised, open-label, phase 3 non-inferiority trial. Lancet. 2012 May 12;379(9828):1791-9. doi: 10.1016/S0140-6736(11)61940-5. Epub 2012 Apr 4. PMID 22480758
- [Background] Kluge R, Chavdarova L, Hoffmann M, Kobe C, Malkowski B, Montravers F, Kurch L, Georgi T, Dietlein M, Wallace WH, Karlen J, Fernandez-Teijeiro A, Cepelova M, Wilson L, Bergstraesser E, Sabri O, Mauz-Korholz C, Korholz D, Hasenclever D. Inter-Reader Reliability of Early FDG-PET/CT Response Assessment Using the Deauville Scale after 2 Cycles of Intensive Chemotherapy (OEPA) in Hodgkin's Lymphoma. PLoS One. 2016 Mar 10;11(3):e0149072. doi: 10.1371/journal.pone.0149072. eCollection 2016. PMID 26963909
- [Background] Hasenclever D, Kurch L, Mauz-Korholz C, Elsner A, Georgi T, Wallace H, Landman-Parker J, Moryl-Bujakowska A, Cepelova M, Karlen J, Alvarez Fernandez-Teijeiro A, Attarbaschi A, Fossa A, Pears J, Hraskova A, Bergstrasser E, Beishuizen A, Uyttebroeck A, Schomerus E, Sabri O, Korholz D, Kluge R. qPET - a quantitative extension of the Deauville scale to assess response in interim FDG-PET scans in lymphoma. Eur J Nucl Med Mol Imaging. 2014 Jul;41(7):1301-8. doi: 10.1007/s00259-014-2715-9. Epub 2014 Mar 7. PMID 24604592
- [Background] Trippett TM, Schwartz CL, Guillerman RP, Gamis AS, Gardner S, Hogan S, London WB, Chen L, de Alarcon P. Ifosfamide and vinorelbine is an effective reinduction regimen in children with refractory/relapsed Hodgkin lymphoma, AHOD00P1: a children's oncology group report. Pediatr Blood Cancer. 2015 Jan;62(1):60-4. doi: 10.1002/pbc.25205. Epub 2014 Oct 12. PMID 25308760
- [Background] Tebbi CK, Mendenhall NP, London WB, Williams JL, Hutchison RE, Fitzgerald TJ, de Alarcon PA, Schwartz C, Chauvenet A. Response-dependent and reduced treatment in lower risk Hodgkin lymphoma in children and adolescents, results of P9426: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2012 Dec 15;59(7):1259-65. doi: 10.1002/pbc.24279. Epub 2012 Aug 21. PMID 22911615